CLINICAL TRIAL: NCT01213784
Title: Optimized Glycemic Control in Type 2 Diabetics With Heart Failure:"Effect on Left Ventricular Function and Skeletal Muscle"
Brief Title: Optimized Glycemic Control in Heart Failure Patients With DM2:"Effect on Left Ventricular Function and Skeletal Muscle"
Acronym: HFDM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M20090047
Record Dates: First submitted 2010-08-24; First posted 2010-10-04 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- optimized diabetic control (Experimental): each participant will be assigned to be optimized in a dedicated diabetic clinic
  Interventions: Other: all antidiabetic drugs will be appliable
- control (No Intervention): participants will be assigned to follow what ever control they were in before the study and not to change any antidiabetic treatment during the interventions period.

INTERVENTIONS:
Other: all antidiabetic drugs will be appliable — We expect all participants to be set on insulin during the intervention, however all types of insulin and other antidiabetics can be used goal: Hba1c lower than 7,5%
  Arms: optimized diabetic control

SUMMARY:
The investigators wish to investigate wether a more strict diabetic control improves cardiac function, muscle strength, exercise capacity and decreases symptoms.

The investigators hypothesis is that improving the glycemic control in suboptimized diabetics with heart failure will improve cardiac performance, muscle strength, exercise capacity and decrease symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction =<45%
* Diabetes
* Hba1c =>7,5%
* In anticongestive treatment
* NYHA class 2-4

Exclusion Criteria:

* Severe angina (CCS 3-4)
* Hemodynamic significant heart valve disease
* Congenital heart disease
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Left ventricular function | 4 month
  Left ventricular function will be evaluated using echocardiografi measuring:
  - 2D Ejection fraction (using an ultrasound agent), global and regional tissue velocity, Strain / strain rate - all measures done during rest and dobutamin stress test.

SECONDARY OUTCOMES:
hormonal and metabolic profile | 4 month
  bloodsamples
6-minutes hall walk test | 4 month
  using a hall walk protocol
Exercise capacity and peak oxygen consumption | 4 month
  using a treadmill test and continues oxygen consumption measurement
Muscle strength and mass | 4 month
  muscle strength: hand grip test

CONTACTS AND LOCATIONS:
Overall Officials: Roni R Nielsen, MD, Principal Investigator — Dept. of cardiology, University hospital Aarhus Skejby
Locations (1):
- Dept. of cardiology, Aarhus university hospital Skejby, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Nielsen R, Wiggers H, Thomsen HH, Bovin A, Refsgaard J, Abrahamsen J, Moller N, Botker HE, Norrelund H. Effect of tighter glycemic control on cardiac function, exercise capacity, and muscle strength in heart failure patients with type 2 diabetes: a randomized study. BMJ Open Diabetes Res Care. 2016 Apr 29;4(1):e000202. doi: 10.1136/bmjdrc-2016-000202. eCollection 2016. PMID 27158520